CLINICAL TRIAL: NCT00503737
Title: Pilot Study of the National Colorectal Cancer Roundtable Toolbox (NCCRT) to Increase Colorectal Cancer Screening Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 25737
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Colorectal Cancer Screening
Keywords: colorectal cancer screening; National Colorectal Cancer Roundtable Toolbox

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colorectal Cancer Screening Toolkit (Active Comparator): Toolbox includes tools and guides designed increase screening by primary care physicians
  Interventions: Behavioral: National Colorectal Cancer Roundtable Toolbox
- Standard of Care Colorectal Cancer Screening (No Intervention): Primary Care physician will screen for colorectal cancer as per his/her standard practice

INTERVENTIONS:
Behavioral: National Colorectal Cancer Roundtable Toolbox
  Arms: Colorectal Cancer Screening Toolkit

SUMMARY:
The American Cancer Society and The Centers for Disease Control and Prevention in collaboration with The National Colorectal Cancer Roundtable published "How to Increase Colorectal Cancer Screening rates in Practice: A Primary Care Clinician's Evidence-Based Toolbox and Guide" in 2005. This toolbox outlines evidence-based interventions aimed at increasing colorectal cancer screening by primary care providers and their office staff. The Toolbox contains the tools to design a multifaceted intervention to increase primary care physician rates of colorectal cancer screening (CRCS). This is a pilot study to look at implementing the toolbox and its affects.

DETAILED DESCRIPTION:
The specific aims of the intervention are: (1) To increase the knowledge of primary care providers as it pertains to current guidelines and communication strategies about colorectal cancer screening (CRCS); (2) To assist offices design a colorectal cancer screening policy, (3) To assist offices adopt a colorectal cancer reminder system and (4) To increase the screening rates of CRC screening. A secondary aim of this project is to synthesize information about the strengths and weaknesses of the toolbox from the primary care physician's (PCP) point of view to aid in future development of an interactive, web-based version of the Toolbox. Our hypothesis is that the practices that implement the toolbox will have a higher rate of colorectal cancer screening than the control group and physician knowledge about CRCS will be increased.

Two of the three sites will be randomly chosen by a number generator to be the intervention sites using the toolbox; the third will be used as a control site. Primary care providers will be defined as Family Practice physicians, General Internists, Nurse Practitioners, and Physician Assistants. Each site has on average of 5-12 providers.

Measurements of baseline rates of CRCS will be assessed by HIPAA compliant chart review for participating providers in the practice by our research coordinator. A list of qualifying patients will be generated by our billing department based on time seen, and billing code. These charts will then be randomly pulled and reviewed by our research coordinator to determine the percentage of eligible subjects who were screened for colorectal cancer (CRC) at each site. A total of 300 charts will be reviewed, broken down into 150 charts pre intervention and 150 charts post intervention. The post intervention chart review will be done at 1 year so that the patients can complete CRCS. The chart review will be done per site (i.e. no link between the individual providers and the patient will be made.) Also the sites will be de-identified so that there is no physician, or group of physicians who are held up to scrutiny.

CRC screening will be considered complete if one of the following was done: (1) Fecal occult blood test (FOBT) in the past year, (2) flexible sigmoidoscopy in the past 5 years, (3) FOBT in the past year and flexible sigmoidoscopy in the past five years (4) double contrast barium enema in the past five years, or (5) colonoscopy in the past 10 years. This will serve as a baseline-screening rate for each practice. Recordable data will be as follows: Sex, Race, Age, Site, Did provider recommend CRCS?, Did the subject follow through with recommendation?, If so, what was the chosen screening modality?, Does the subject have a family history of a 1st or 2nd degree relative with CRC?, Does the subject have a family history of a 1st or 2nd degree relative with adenomatous polyps? For the providers in the intervention group, they will be asked to attend a lunchtime lecture given by the PI on CRCS. They will also be asked to do a 20 question pre and post intervention questionnaire and a pre and post intervention health care provider survey. They will also be provided with brochures from the American Cancer Society. The providers in the control group will only complete the survey and the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Health care providers who are currently practicing and recommending CRCS.

Exclusion Criteria:

* Any provider not at the clinics of interest

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 287 (Actual)
Dates: Start 2007-09; Primary Completion 2010-09-01 (Actual); Study Completion 2010-09-01 (Actual)

PRIMARY OUTCOMES:
Increase the knowledge of providers as it pertains to current guidelines and strategies about CRCS; assist offices design a CRCS policy, assist offices adopt a CRC reminder system and increase the screening rates of CRC. | 2 years

SECONDARY OUTCOMES:
synthesize information about the strengths and weaknesses of the toolbox from the primary care physician's (PCP) point of view to aid in future development of an interactive, web-based version of the Toolbox. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Downey, MD, Principal Investigator — Penn State College of Medicine, Penn State Milton S. Hershey Medical Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States